CLINICAL TRIAL: NCT03582267
Title: The Effect of Docosahexaenoic Acid Supplementation on Biomarkers of Concussion Over the Course of a Year in Canadian National Rugby Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Christian University (Other)
Responsible Party: Principal Investigator, Jonathan Oliver, Assistant Professor, Texas Christian University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 1706-066-1706
Record Dates: First submitted 2018-06-27; First posted 2018-07-10 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Head Trauma
MeSH Terms: conditions — Craniocerebral Trauma | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary Supplement (Experimental): Docosahexaenoic Acid (DHA)
  Interventions: Dietary Supplement: Docosahexaenoic Acid (DHA)
- No Intervention (No Intervention): No Docosahexaenoic Acid supplementation

INTERVENTIONS:
Dietary Supplement: Docosahexaenoic Acid (DHA) — Daily administration of docosahexaenoic Acid (DHA). 2 grams of DHA liquid concentrate administered per day throughout trial period.
  Other Names: Brain Armor DHA Liquid Concentrate
  Arms: Dietary Supplement

SUMMARY:
Nutrition interventions may present a safe and relatively risk free intervention for protection against subconcussive impacts. Docosahexaenoic acid (DHA, 22:6n-3) is the principal Omega 3 polyunsaturated fatty acid in the brain, playing an integral role in the brain's development and structural integrity. The goal of this study is to determine if supplementation with DHA attenuates blood biomarkers of repetitive head trauma linked to sub-concussive impacts sustained in rugby participation.

ELIGIBILITY:
Inclusion Criteria:

* Canadian national rugby athletes on 7s and 15s teams

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Blood concentration of neurofilament light protein | 12 times throughout course of 1 year
  Concentrations of neuronally derived proteins measured in blood

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Christian Universti, Fort Worth, Texas, United States